CLINICAL TRIAL: NCT06084351
Title: Phase 3 Open-Label Controlled Trial of Convalescent Plasma in Early COVID-19 Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCH- 1Apr2020
Record Dates: First submitted 2020-07-22; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental)
  Interventions: Drug: Convalescent Plasma
- Standard of care (Active Comparator)
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Convalescent Plasma — Class: Blood product Physical Description: Opaque yellow fluid within a container labelled with the statement "Caution: New Drug - Limited by Federal (or United States) law to investigational use)." Container will also be labelled with the International Society of Blood Transfusion format for Blood Components. Label will contain the expiration date and the donor identification number. Label will also contain information pertaining to the ABO typing of the plasma. A copy of the IBST identifier will be placed with the patient chart.
  Manufacture: Plasma will be collected via apheresis via collaboration with American Blood Bank Corporation, a FDA-registered blood establishment. The donors will be screened in accordance with the FDA guidance for donor eligibility for COVID-19:
  Arms: Convalescent Plasma
Other: Standard of Care — Standard of care treatment for hospitalized COVID-19 patients
  Arms: Standard of care

SUMMARY:
The expanded access program for investigational convalescent plasma (CP) is being utilized nationwide despite its unproven benefit and optimal timing of transfusion. The optimal administration of CP during a viral pandemic must consider the supply of the product, ideal patient selection, and appropriate timing in order to produce maximum benefit with a scarce resource [2]. Currently, the FDA suggested guidelines for use include "severe", "critical" or at risk for critical disease. The optimal administration of CP with anti-SARS-CoV-2 antibodies is theoretically early in the course of the illness [1], before multiorgan failure or a maladaptive immune response, like seen in the cytokine release syndrome, occurs. Our open-label trial will randomize COVID-19+ patients admitted to the hospital who are at high risk for severe disease to receive 1 dose CP ordered within 48 hours of admission plus standard of care vs. standard of care. The primary clinical endpoint will be time to clinical improvement within 28 days after randomization (based on the ordinal scale as specified below). The purpose of this trial will be to obtain data which can be further utilized in future clinical trials and help clinicians understand the effectiveness of CP.

DETAILED DESCRIPTION:
Based on previous veterinary and human studies of coronavirus vaccines, it is probable that an effective vaccine is 1-2 years away. Multiple antiviral medications are being currently studied, but manufacturing capacity of adequate quantities may be 6-12 months away from the identification of an effective drug. In addition, effective drugs or a vaccine may not be available to all countries given current international shortages. Conversely, blood banks have a well established infrastructure for the collection and distribution of convalescent plasma. If convalescent plasma is effective in the treatment of COVID-19, it would be accessible much more quickly, and would likely be available in all geopolitical regions and all economic strata. Therefore, it is imperative to study all possible approaches to the use of convalescent plasma. Based on other antiviral therapies, and previous experience with convalescent plasma, we believe it is very likely that early use of plasma will be more likely to be effective as therapy in COVID-19. Our study is designed to explore the possibility that early use is beneficial.

Convalescent plasma has been used successfully in previous viral outbreaks, including 1918 influenza pandemic, MERS, previous SARS, Ebola virus and others. The goal of this study is to provide rapid data the medical community can use to evaluate its effectiveness in the current pandemic.

The current FDA emergency authorization for CP allows for its use in severe, critical or at risk for critical disease as defined by the FDAs suggested guidelines for use. It has been documented that some of the mortality and morbidity associated with COVID-19 is related to the cytokine release syndrome due to an overactivated immune response. The theoretical optimal time for convalescent plasma infusion is early in the course, when viremia peaks and the primary immune response has yet to adequately suppress the viral illness [1]. Scarce resources during pandemics should be utilized to achieve maximum benefit [2]. We are proposing a study which aims to document early intervention in a high risk group. Once this information is available, and if it is found to be effective, we believe COVID-19 recovered patients will be easier to recruit into other "from community to community" plasma donation systems such as ours.

1. After informed consent is obtained, the enrolling physician will be required to present the case to the principal investigator to ensure they meet inclusion criteria. The trial sponsor Larkin Community Hospital has published internal protocols pertaining to the recommended laboratory monitoring for COVID-19 patients which should be followed by all physicians enrolling patients in the trial; these guidelines include: D-dimer, C-reactive protein, lactate dehydrogenase, and ferritin level (at admission and every 48 hours), complete blood count and comprehrensive metabolic panel (at admission and daily); and electrocardiogram and chest x-ray (at admission and with changes in clinical status). Arterial blood gas will be ordered for any Intensive Care admission or at attending physician's discretion.
2. After obtaining patient consent, patients will be assigned a study ID which will correlate to the patient's medical record. The list with patient identifiers will be held only by the investigative team. The ordering physician will not know to which group the patient will be assigned until after enrollment. Patients will be stratified by age at time of enrollment (40-64 years old, 65-79 years, 80+ years). The stratified patients will then be randomized using variable block sizes using an electronically generated randomization scheme (e.g. www.randomization.com) to either the convalescent plasma treatment group or standard care.

4. Patients in the treatment arm will receive 1 unit (minimum 200mL) of ABO compatible convalescent plasma one time. ABO compatible convalescent plasma units will be obtained from a registered or licensed blood collector following registration of the patient.

5. ABO compatible COVID-19 CP will be administered according to standard hospital procedures and in accordance with the FDA guidance on use of convalescent plasma. For practical purposes, one unit of ABO compatible CP will be administered. This will be provided by a registered or licensed blood collector and will be collected by apheresis. Pre-infusion acetaminophen (IV, PO, via PEG/nasogastric tube, Rectal) and/or diphenhydramine (PO, IV, via PEG/nasogastric tube) at the discretion of the attending physician. The duration of infusion will usually take 1 to 2 hours (rate of 100 to 200 mL/hr).

6. COVID-19 CP will be supplied as an investigational blood product for the treatment of COVID-19 with either a label or tie tag on the bag indicating the presence of COVID-19 antibodies. The licensed or registered blood collector will follow the Circular of Information and FDA's regulations and the additional considerations for convalescent plasma on the FDA's webpage (https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/recommendations-investigational-covid-19-convalescent-plasma). Local institutional guidelines for conventional plasma administration will be followed prior to administration including ABO compatibility checks and thawing. Monitoring for transfusion reactions will occur the same as for standard blood product infusion. It should be noted, currently 1 retention sample of frozen whole blood will be kept for study in the future regarding antibody titers should it become available at our institution. The study may at some point require minimum titers of antibody in the blood product to be considered for use (1:160) 7. The study involves the one-time administration of ABO matched COVID-19 CP, and patients are free to withdraw consent from participation at any time.

8. In the event of minor transfusion reactions, the transfusion will continue as planned with medication to mitigate the reaction (e.g. diphenhydramine for pruritis). If the patient is unable to tolerate continued transfusion despite medication, the transfusion will be halted. If there are any indications of a severe or systemic transfusion reaction, the transfusion will be halted immediately, and an investigation will be performed by the trial sponsor to identify and classify the type of reaction (e.g. TRALI v. anaphylactoid reaction v. acute hemolytic reaction) as well as to ensure proper procedure was maintained (e.g. ABO typing and confirmation; appropriate infusion rate, appropriate patient monitoring during infusion).

9. Patients' will be followed in the study until discharge, 28 days after enrollment, withdrawal of consent from trial, or death: whichever happens earliest. Adverse events, including but not limited to: transfusion reactions and adverse clinical outcomes will be reported to the trial sponsor and IRB. The trial sponsor will investigate any adverse events to determine if they may be related to the investigational drug. If an adverse event is deemed to be reportable, it will be reported via the FDA Adverse Event Reporting System (FDAERS) (in no more than 7 days in the case of severe/life-threatening cases and in no more than 15 days in the case of any adverse event).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the participating acute care facilities as listed above (Larkin Palm Springs Hospital, Larkin South Miami Hospital) AND enrolled in the trial within 48 hours of hospital admission (defined by when admission order was placed) AND
* Age ≥ 40 with at least one of the following comorbidities (hypertension, diabetes mellitus, coronary artery disease, congestive heart failure, pulmonary hypertension, idiopathic pulmonary fibrosis, asthma, COPD, cancer, HIV/AIDS, chronic kidney disease, immunosuppression, obesity). OR
* Age ≥ 65 years of age with or without comorbid conditions. AND
* Severe or life-threatening COVID-19 disease as defined by the FDA:
* "Severe disease is defined as one or more of the following: shortness of breath (dyspnea), respiratory frequency ≥ 30/min, blood oxygen saturation ≤ 93%, partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300, lung infiltrates > 50% within 24 to 48 hours, Life-threatening disease is defined as one or more of the following: respiratory failure, septic shock, multiple organ dysfunction or failure AND
* Positive COVID-19 test via nasopharyngeal or pharyngeal PCR.
* Able to consent to treatment

Exclusion Criteria:

* Unable to consent
* Lack of laboratory confirmed COVID-19 infection.
* Hospice/Palliative care
* Unable to tolerate 200mL of fluid.
* History of IgA deficiency (due to risk of reaction)
* History of anaphylactoid or other severe reaction to plasma or blood products.
* Philosophical/Religious objections to receiving blood products.
* Pregnant or breastfeeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical Improvement within 28 days of randomization | 7, 14 and 28 days after randomization
  Clinical improvement will be defined as a two-point reduction in patients' admission status on a 6-point ordinal scale, or discharge from the hospital, whichever comes first. The 6-point scale is as follows:
  Discharged = 0 Not requiring supplemental oxygen =1 Requiring supplemental oxygen =2 Requiring noninvasive mechanical ventilation =3 Requiring invasive mechanical ventilation = 4 Death = 5

SECONDARY OUTCOMES:
Mortality at day 28; frequency of invasive mechanical ventilation; duration of oxygen therapy; duration of hospital admission | Within 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Larkin Community Hospital, South Miami, Florida, United States

REFERENCES:
- [Background] Russell CD, Millar JE, Baillie JK. Clinical evidence does not support corticosteroid treatment for 2019-nCoV lung injury. Lancet. 2020 Feb 15;395(10223):473-475. doi: 10.1016/S0140-6736(20)30317-2. Epub 2020 Feb 7. No abstract available. PMID 32043983
- [Result] Emanuel EJ, Persad G, Upshur R, Thome B, Parker M, Glickman A, Zhang C, Boyle C, Smith M, Phillips JP. Fair Allocation of Scarce Medical Resources in the Time of Covid-19. N Engl J Med. 2020 May 21;382(21):2049-2055. doi: 10.1056/NEJMsb2005114. Epub 2020 Mar 23. No abstract available. PMID 32202722